CLINICAL TRIAL: NCT00321620
Title: A Randomized, Double-Blind, Multicenter Study of Denosumab Compared With Zoledronic Acid (Zometa®) in the Treatment of Bone Metastases in Men With Hormone-Refractory Prostate Cancer
Brief Title: Study of Denosumab vs. Zoledronic Acid to Treat Bone Metastases in Men With Hormone-refractory Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 20050103
Record Dates: First submitted 2006-05-02; First posted 2006-05-04 (Estimated); Results first posted 2014-03-21 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Bone Metastases
Keywords: Bone metastases; Hormone-refractory prostate cancer; Skeletal; Fractures; Compressions; Bisphosphonates
MeSH Terms: conditions — Fractures, Bone | interventions — Zoledronic Acid; Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zoledronic acid (Active Comparator)
  Interventions: Drug: zoledronic acid
- denosumab (Experimental)
  Interventions: Biological: denosumab

INTERVENTIONS:
Drug: zoledronic acid — Q4W 4 mg zoledronic acid IV over minimum 15 minutes and 120 mg denosumab placebo SC
  Other Names: Zometa
  Arms: zoledronic acid
Biological: denosumab — Q4W 120 mg denosumab SC and 4 mg zoledronic acid placebo IV over a minimum of 15 minutes
  Arms: denosumab

SUMMARY:
The purpose of this study is to determine if denosumab is non-inferior to zoledronic acid (Zometa®) in the treatment of bone metastases in men with hormone-refractory prostate cancer

ELIGIBILITY:
Inclusion Criteria:

* Men >/= 18 years of age with histologically confirmed prostate cancer
* Radiographic evidence of at least one bone metastasis
* Failure of at least one hormonal therapy as evidenced by a rising PSA
* Serum testosterone level of <50 ng/dL
* ECOG PS 0, 1, or 2
* Adequate organ function

Exclusion Criteria:

* Current or prior IV bisphosphonate administration
* Current or prior oral bisphosphonates for bone mets
* Life expectancy of less than 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1904 (Actual)
Dates: Start 2006-04-01 (Actual); Primary Completion 2009-10-01 (Actual); Study Completion 2012-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Fizazi K, Carducci M, Smith M, Damiao R, Brown J, Karsh L, Milecki P, Shore N, Rader M, Wang H, Jiang Q, Tadros S, Dansey R, Goessl C. Denosumab versus zoledronic acid for treatment of bone metastases in men with castration-resistant prostate cancer: a randomised, double-blind study. Lancet. 2011 Mar 5;377(9768):813-22. doi: 10.1016/S0140-6736(10)62344-6. Epub 2011 Feb 25. PMID 21353695
- [Background] Smith MR, Coleman RE, Klotz L, Pittman K, Milecki P, Ng S, Chi KN, Balakumaran A, Wei R, Wang H, Braun A, Fizazi K. Denosumab for the prevention of skeletal complications in metastatic castration-resistant prostate cancer: comparison of skeletal-related events and symptomatic skeletal events. Ann Oncol. 2015 Feb;26(2):368-74. doi: 10.1093/annonc/mdu519. Epub 2014 Nov 25. PMID 25425475
- [Background] Fizazi K, Massard C, Smith M, Rader M, Brown J, Milecki P, Shore N, Oudard S, Karsh L, Carducci M, Damiao R, Wang H, Ying W, Goessl C. Bone-related Parameters are the Main Prognostic Factors for Overall Survival in Men with Bone Metastases from Castration-resistant Prostate Cancer. Eur Urol. 2015 Jul;68(1):42-50. doi: 10.1016/j.eururo.2014.10.001. Epub 2014 Oct 29. PMID 25449207
- [Derived] Jakob T, Tesfamariam YM, Macherey S, Kuhr K, Adams A, Monsef I, Heidenreich A, Skoetz N. Bisphosphonates or RANK-ligand-inhibitors for men with prostate cancer and bone metastases: a network meta-analysis. Cochrane Database Syst Rev. 2020 Dec 3;12(12):CD013020. doi: 10.1002/14651858.CD013020.pub2. PMID 33270906
- [Derived] Stopeck AT, Fizazi K, Body JJ, Brown JE, Carducci M, Diel I, Fujiwara Y, Martin M, Paterson A, Tonkin K, Shore N, Sieber P, Kueppers F, Karsh L, Yardley D, Wang H, Maniar T, Arellano J, Braun A. Safety of long-term denosumab therapy: results from the open label extension phase of two phase 3 studies in patients with metastatic breast and prostate cancer. Support Care Cancer. 2016 Jan;24(1):447-455. doi: 10.1007/s00520-015-2904-5. Epub 2015 Sep 3. PMID 26335402
- [Derived] Body JJ, Bone HG, de Boer RH, Stopeck A, Van Poznak C, Damiao R, Fizazi K, Henry DH, Ibrahim T, Lipton A, Saad F, Shore N, Takano T, Shaywitz AJ, Wang H, Bracco OL, Braun A, Kostenuik PJ. Hypocalcaemia in patients with metastatic bone disease treated with denosumab. Eur J Cancer. 2015 Sep;51(13):1812-21. doi: 10.1016/j.ejca.2015.05.016. Epub 2015 Jun 17. PMID 26093811
- [Derived] de Liano AG, Reig O, Mellado B, Martin C, Rull EU, Maroto JP. Prognostic and predictive value of plasma testosterone levels in patients receiving first-line chemotherapy for metastatic castrate-resistant prostate cancer. Br J Cancer. 2014 Apr 29;110(9):2201-8. doi: 10.1038/bjc.2014.189. Epub 2014 Apr 10. PMID 24722180
- [Derived] von Moos R, Body JJ, Egerdie B, Stopeck A, Brown JE, Damyanov D, Fallowfield LJ, Marx G, Cleeland CS, Patrick DL, Palazzo FG, Qian Y, Braun A, Chung K. Pain and health-related quality of life in patients with advanced solid tumours and bone metastases: integrated results from three randomized, double-blind studies of denosumab and zoledronic acid. Support Care Cancer. 2013 Dec;21(12):3497-507. doi: 10.1007/s00520-013-1932-2. Epub 2013 Aug 22. PMID 23975226
- [Derived] Lipton A, Fizazi K, Stopeck AT, Henry DH, Brown JE, Yardley DA, Richardson GE, Siena S, Maroto P, Clemens M, Bilynskyy B, Charu V, Beuzeboc P, Rader M, Viniegra M, Saad F, Ke C, Braun A, Jun S. Superiority of denosumab to zoledronic acid for prevention of skeletal-related events: a combined analysis of 3 pivotal, randomised, phase 3 trials. Eur J Cancer. 2012 Nov;48(16):3082-92. doi: 10.1016/j.ejca.2012.08.002. Epub 2012 Sep 10. PMID 22975218
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 12 May 2006 through 18 December 2008.
Pre-assignment Details: 1904 participants were enrolled, however 3 were excluded from all analyses as Institutional Review Board review activities and oversight were not ensured.
Groups:
- Zoledronic Acid: Zoledronic acid 4 mg by intravenous injection with a subcutaneous denosumab placebo once every 4 weeks
- Denosumab: Denosumab 120 mg subcutaneously with an intravenous zoledronic acid placebo once every 4 weeks
Period: Overall Study
Arm/Group | Zoledronic Acid | Denosumab
Started | 951 | 950
Received Investigational Product | 946 | 942
Completed | 208 | 228
Not Completed | 743 | 722
Not completed — Death | 269 | 294
Not completed — Withdrawal by Subject | 164 | 147
Not completed — Disease progression | 113 | 117
Not completed — Adverse Event | 43 | 56
Not completed — Lost to Follow-up | 13 | 9
Not completed — Physician Decision | 4 | 1
Not completed — Noncompliance | 14 | 7
Not completed — Protocol deviation | 4 | 3
Not completed — Ineligibility determined | 2 | 3
Not completed — Participant request | 75 | 52
Not completed — Other | 42 | 33

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | Denosumab | Total
Number analyzed (Participants) | 951 | 950 | 1901
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.0 (8.4) | 70.5 (8.7) | 70.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 951 | 950 | 1901
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 810 | 829 | 1639
  Black or African American | 35 | 38 | 73
  Hispanic or Latino | 57 | 45 | 102
  Asian | 26 | 22 | 48
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Other | 22 | 15 | 37
Prostate-Specific Antigen (PSA) Stratification Factor [Number; unit: Participants]
  PSA level < 10 ng/mL | 145 | 145 | 290
  PSA level ≥ 10 ng/mL | 806 | 805 | 1611
Previous Skeletal-Related Event (SRE) Stratification Factor [Number; unit: Participants]
  Yes | 231 | 232 | 463
  No | 720 | 718 | 1438
Current Prostate Cancer Chemotherapy Stratification Factor [Number; unit: Participants] — Defined as within 6 weeks before randomization
  Participants
    Yes | 132 | 132 | 264
    No | 819 | 818 | 1637

OUTCOME MEASURES:

1. Primary Outcome: Time to the First On-Study SRE (Non-inferiority)
Description: Time to the first on-study skeletal-related event (SRE) analyzed for non-inferiority. Kaplan-Meier estimates of the median and its dispersion are reported.
Time Frame: Up to 40.5 months
Population: Full Analysis Set, composed of all randomized participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 951 | 950
Days | 521.0 [456.00 to 592.00] | 629.0 [573.00 to 757.00]
Statistical Analysis 1: Comparison: Zoledronic Acid vs Denosumab; Test type: Non-Inferiority or Equivalence — A synthesis method was used for the non-inferiority test for the hypothesis that denosumab preserves as least 50% of the effect of zoledronic acid vs. placebo; p = 0.0002, Regression, Cox; Hazard Ratio (HR) = 0.82, 95% CI [0.71 to 0.95] — Stratified by the randomization stratification factors (previous skeletal-related event, prostate-specific antigen level, and current chemotherapy)

2. Secondary Outcome: Time to the First On-Study SRE (Superiority)
Description: Time to the first on-study skeletal-related event (SRE), analyzed for superiority of denosumab. Kaplan-Meier estimates of the median and its dispersion are reported.
Time Frame: Up to 40.5 months
Population: Full Analysis Set, composed of all randomized participants
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 951 | 950
Days | 521.0 [456.0 to 592.0] | 629.0 [573.00 to 757.00]
Statistical Analysis 1: Comparison: Zoledronic Acid vs Denosumab; Test type: Superiority or Other; p = 0.0085, Regression, Cox; P-value was adjusted for multiplicity according to a hierarchical testing strategy and Hochberg procedure; Hazard Ratio (HR) = 0.82, 95% CI [0.71 to 0.95] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Time to the First-And-Subsequent On-Study SRE
Description: Time to the first-and-subsequent on-study skeletal-related event (SRE), analyzed for superiority of denosumab using multiple event analysis, the event must occur at least 21 days after the previous SRE.
  This outcome measure utilizes multiple event times, was analyzed based on a proportional mean model, and is therefore more appropriately summarized by the cumulative mean number of events.
Time Frame: Up to 40.5 months
Population: Full Analysis Set, composed of all randomized participants
Measure: Number; unit: Events
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 951 | 950
Events | 584 | 494
Statistical Analysis 1: Comparison: Zoledronic Acid vs Denosumab; Test type: Superiority or Other; p = 0.0085, Anderson-Gill model; P-value was adjusted for multiplicity according to a hierarchical testing strategy and Hochberg procedure; Rate ratio = 0.82, 95% CI [0.71 to 0.94] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: up to 3 years 5 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
  One subject who was randomized to zoledronic acid and received denosumab as the 1st investigational product was analyzed on the denosumab arm for safety analyses.
Arm/Group | Zoledronic Acid 4 mg Q4W | Denosumab 120 mg Q4W
Serious Adverse Events (participants affected / at risk) | 568/945 | 594/943
Other Adverse Events (participants affected / at risk) | 853/945 | 844/943
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 4 mg Q4W (N=945) | Denosumab 120 mg Q4W (N=943)
Anaemia (Blood and lymphatic system disorders) | 82 | 108
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 3
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 8
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 4 | 10
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 3 | 1
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 10
Acute coronary syndrome (Cardiac disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 7 | 5
Angina pectoris (Cardiac disorders) | 5 | 1
Angina unstable (Cardiac disorders) | 1 | 2
Arrhythmia (Cardiac disorders) | 2 | 6
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 8 | 10
Atrial flutter (Cardiac disorders) | 3 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bundle branch block right (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 4 | 5
Cardiac asthma (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 23 | 21
Cardiac failure acute (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 7 | 8
Cardio-respiratory arrest (Cardiac disorders) | 12 | 7
Cardiogenic shock (Cardiac disorders) | 0 | 2
Cardiomegaly (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 6 | 2
Cardiovascular insufficiency (Cardiac disorders) | 3 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 2 | 2
Myocardial infarction (Cardiac disorders) | 13 | 9
Myocardial ischaemia (Cardiac disorders) | 6 | 5
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 2
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 3
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Acute vestibular syndrome (Ear and labyrinth disorders) | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Blindness unilateral (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 3
Retinal artery thrombosis (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 12 | 8
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 3
Anal fissure (Gastrointestinal disorders) | 0 | 2
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 2
Colitis (Gastrointestinal disorders) | 1 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 9 | 5
Diarrhoea (Gastrointestinal disorders) | 13 | 12
Dysphagia (Gastrointestinal disorders) | 1 | 2
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 2 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 3
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 2
Gingival bleeding (Gastrointestinal disorders) | 0 | 2
Haematemesis (Gastrointestinal disorders) | 3 | 2
Haematochezia (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 3
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 0
Intestinal obstruction (Gastrointestinal disorders) | 4 | 4
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 14 | 8
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 2
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 3
Rectal stenosis (Gastrointestinal disorders) | 1 | 0
Rectourethral fistula (Gastrointestinal disorders) | 0 | 1
Reflux gastritis (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 3
Stomatitis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 6
Vomiting (Gastrointestinal disorders) | 22 | 24
Abasia (General disorders) | 1 | 0
Asthenia (General disorders) | 29 | 37
Catheter related complication (General disorders) | 3 | 2
Catheter site pain (General disorders) | 1 | 1
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 13 | 9
Chills (General disorders) | 1 | 0
Death (General disorders) | 10 | 11
Discomfort (General disorders) | 1 | 0
Disease progression (General disorders) | 2 | 0
Drug intolerance (General disorders) | 1 | 0
Fatigue (General disorders) | 10 | 20
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 28 | 29
Generalised oedema (General disorders) | 1 | 2
Hernia (General disorders) | 0 | 1
Impaired healing (General disorders) | 0 | 1
Inflammation (General disorders) | 0 | 1
Localised oedema (General disorders) | 2 | 0
Malaise (General disorders) | 3 | 3
Mucosal inflammation (General disorders) | 2 | 0
Multi-organ failure (General disorders) | 18 | 18
Oedema (General disorders) | 3 | 1
Oedema peripheral (General disorders) | 8 | 13
Pain (General disorders) | 12 | 16
Performance status decreased (General disorders) | 2 | 9
Pyrexia (General disorders) | 18 | 19
Sudden death (General disorders) | 2 | 3
Suprapubic pain (General disorders) | 1 | 0
Terminal state (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 3 | 0
Cholelithiasis obstructive (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 6 | 10
Hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Abscess intestinal (Infections and infestations) | 0 | 1
Alveolar osteitis (Infections and infestations) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Bacteraemia (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 6
Bronchopneumonia (Infections and infestations) | 1 | 3
Candidiasis (Infections and infestations) | 0 | 1
Catheter related infection (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 4 | 6
Central line infection (Infections and infestations) | 1 | 0
Cholecystitis infective (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Dermo-hypodermitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 1
Endotoxaemia (Infections and infestations) | 0 | 1
Enterococcal sepsis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 1 | 2
Fungal oesophagitis (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 3 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal infection (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 2 | 1
Infection (Infections and infestations) | 3 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 3
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Ludwig angina (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 3 | 2
Meningitis bacterial (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 2 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 3
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 0 | 1
Penile abscess (Infections and infestations) | 1 | 0
Peridiverticulitis (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 24 | 40
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 0
Post procedural sepsis (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 2 | 4
Pyelonephritis acute (Infections and infestations) | 1 | 2
Pyelonephritis chronic (Infections and infestations) | 1 | 1
Renal abscess (Infections and infestations) | 1 | 1
Scrotal abscess (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 11 | 12
Septic shock (Infections and infestations) | 4 | 5
Skin infection (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 3
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tongue abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 30 | 28
Urosepsis (Infections and infestations) | 4 | 5
Wound infection (Infections and infestations) | 0 | 1
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 1 | 0
Device failure (Injury, poisoning and procedural complications) | 1 | 0
Device malfunction (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 2
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 4
Femur fracture (Injury, poisoning and procedural complications) | 3 | 4
Fracture (Injury, poisoning and procedural complications) | 1 | 1
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 3
Ilium fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Kidney rupture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 4 | 0
Medical device discomfort (Injury, poisoning and procedural complications) | 0 | 1
Mouth injury (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Renal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 2 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Stent occlusion (Injury, poisoning and procedural complications) | 0 | 1
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 7
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 3
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Aspiration bronchial (Investigations) | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 1
Blood creatinine (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 0 | 5
Blood pressure systolic abnormal (Investigations) | 0 | 1
Blood urine present (Investigations) | 0 | 1
General physical condition abnormal (Investigations) | 1 | 0
Glomerular filtration rate (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 6 | 2
Hepatic enzyme increased (Investigations) | 0 | 1
International normalised ratio decreased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Occult blood positive (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 2 | 0
Prostatic specific antigen increased (Investigations) | 1 | 4
Prothrombin time prolonged (Investigations) | 0 | 1
Urine output decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 12 | 14
Decreased appetite (Metabolism and nutrition disorders) | 13 | 13
Dehydration (Metabolism and nutrition disorders) | 19 | 36
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 2 | 2
Feeding disorder (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 6
Hypermetabolism (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hyperosmolar state (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 7 | 24
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 6
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 3
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 36 | 29
Bone pain (Musculoskeletal and connective tissue disorders) | 34 | 24
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 9
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4 | 14
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 10
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Sarcopenia (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 10
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 14
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 13
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3
Metastases to rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 56 | 34
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 17 | 8
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Waldenstrom's macroglobulinaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Brown-Sequard syndrome (Nervous system disorders) | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 1 | 0
Cerebral artery embolism (Nervous system disorders) | 1 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 5 | 4
Cerebral infarction (Nervous system disorders) | 0 | 2
Cerebral ischaemia (Nervous system disorders) | 4 | 5
Cerebrovascular accident (Nervous system disorders) | 5 | 15
Cerebrovascular disorder (Nervous system disorders) | 2 | 2
Cervical cord compression (Nervous system disorders) | 1 | 1
Cognitive disorder (Nervous system disorders) | 1 | 1
Convulsion (Nervous system disorders) | 2 | 2
Depressed level of consciousness (Nervous system disorders) | 2 | 0
Diabetic hyperglycaemic coma (Nervous system disorders) | 0 | 1
Diplegia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 3
Dysaesthesia (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Embolic stroke (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 0 | 1
Epidural lipomatosis (Nervous system disorders) | 1 | 0
Facial palsy (Nervous system disorders) | 1 | 3
Facial paresis (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 2
Haemorrhagic stroke (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 4 | 1
Hemiparesis (Nervous system disorders) | 1 | 2
Hemiplegia (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 1
Hypertonia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 2 | 1
Hypotonia (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1
Lethargy (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 2 | 3
Mental impairment (Nervous system disorders) | 0 | 1
Monoparesis (Nervous system disorders) | 2 | 2
Myoclonus (Nervous system disorders) | 1 | 0
Nerve root compression (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 2
Neurological decompensation (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 4 | 1
Paralysis (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 2 | 1
Paraplegia (Nervous system disorders) | 5 | 4
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Radicular syndrome (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 1 | 1
Spinal cord compression (Nervous system disorders) | 33 | 24
Spinal cord ischaemia (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 6 | 10
Transient ischaemic attack (Nervous system disorders) | 4 | 3
Trigeminal neuralgia (Nervous system disorders) | 0 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 2
Confusional state (Psychiatric disorders) | 10 | 12
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 2
Disorientation (Psychiatric disorders) | 2 | 1
Emotional distress (Psychiatric disorders) | 1 | 0
Hypochondriasis (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 2 | 1
Sopor (Psychiatric disorders) | 0 | 1
Anuria (Renal and urinary disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 4 | 1
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Bladder perforation (Renal and urinary disorders) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 1 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 2 | 2
Faecaluria (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 37 | 23
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 3
Hydronephrosis (Renal and urinary disorders) | 12 | 19
Neurogenic bladder (Renal and urinary disorders) | 1 | 0
Obstructive uropathy (Renal and urinary disorders) | 4 | 2
Oliguria (Renal and urinary disorders) | 0 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 2
Polyuria (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1
Renal disorder (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 28 | 26
Renal failure acute (Renal and urinary disorders) | 16 | 18
Renal failure chronic (Renal and urinary disorders) | 2 | 2
Renal impairment (Renal and urinary disorders) | 5 | 2
Renal pain (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 2 | 2
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1
Urethral obstruction (Renal and urinary disorders) | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 1 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 2 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 2
Urinary retention (Renal and urinary disorders) | 35 | 32
Urinary tract disorder (Renal and urinary disorders) | 0 | 3
Urinary tract obstruction (Renal and urinary disorders) | 6 | 5
Urine odour abnormal (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Genital pain (Reproductive system and breast disorders) | 1 | 0
Oedema genital (Reproductive system and breast disorders) | 4 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 1
Penile pain (Reproductive system and breast disorders) | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 1 | 0
Prostatic cyst (Reproductive system and breast disorders) | 1 | 0
Prostatic disorder (Reproductive system and breast disorders) | 0 | 1
Prostatic haemorrhage (Reproductive system and breast disorders) | 1 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 2
Prostatomegaly (Reproductive system and breast disorders) | 2 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 | 36
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 12
Pleural haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 16 | 20
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 | 24
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 0
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Walking disability (Social circumstances) | 1 | 0
Catheter placement (Surgical and medical procedures) | 0 | 1
Ostectomy (Surgical and medical procedures) | 0 | 1
Spinal operation (Surgical and medical procedures) | 1 | 0
Transurethral prostatectomy (Surgical and medical procedures) | 3 | 2
Ureteral stent insertion (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 8 | 8
Embolism (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1
Extrinsic vascular compression (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 5
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 8 | 8
Hypovolaemic shock (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 2 | 0
Phlebitis (Vascular disorders) | 2 | 2
Shock (Vascular disorders) | 1 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 3 | 0
Venous thrombosis (Vascular disorders) | 2 | 2
Venous thrombosis limb (Vascular disorders) | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 4 mg Q4W (N=945) | Denosumab 120 mg Q4W (N=943)
Anaemia (Blood and lymphatic system disorders) | 313 | 300
Abdominal pain (Gastrointestinal disorders) | 57 | 67
Constipation (Gastrointestinal disorders) | 247 | 233
Diarrhoea (Gastrointestinal disorders) | 143 | 174
Nausea (Gastrointestinal disorders) | 242 | 271
Vomiting (Gastrointestinal disorders) | 138 | 155
Asthenia (General disorders) | 226 | 219
Chest pain (General disorders) | 62 | 67
Fatigue (General disorders) | 217 | 247
Oedema peripheral (General disorders) | 171 | 187
Pain (General disorders) | 85 | 78
Pyrexia (General disorders) | 121 | 87
Urinary tract infection (Infections and infestations) | 105 | 88
Blood creatinine increased (Investigations) | 50 | 41
Weight decreased (Investigations) | 131 | 150
Decreased appetite (Metabolism and nutrition disorders) | 263 | 264
Hypocalcaemia (Metabolism and nutrition disorders) | 45 | 105
Arthralgia (Musculoskeletal and connective tissue disorders) | 197 | 188
Back pain (Musculoskeletal and connective tissue disorders) | 271 | 290
Bone pain (Musculoskeletal and connective tissue disorders) | 230 | 221
Muscle spasms (Musculoskeletal and connective tissue disorders) | 27 | 51
Muscular weakness (Musculoskeletal and connective tissue disorders) | 58 | 52
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 54 | 47
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 133 | 111
Myalgia (Musculoskeletal and connective tissue disorders) | 57 | 36
Pain in extremity (Musculoskeletal and connective tissue disorders) | 184 | 192
Dizziness (Nervous system disorders) | 63 | 54
Headache (Nervous system disorders) | 71 | 61
Paraesthesia (Nervous system disorders) | 69 | 53
Anxiety (Psychiatric disorders) | 52 | 45
Depression (Psychiatric disorders) | 39 | 50
Insomnia (Psychiatric disorders) | 94 | 89
Dysuria (Renal and urinary disorders) | 52 | 62
Haematuria (Renal and urinary disorders) | 76 | 76
Urinary retention (Renal and urinary disorders) | 47 | 62
Cough (Respiratory, thoracic and mediastinal disorders) | 82 | 91
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 95 | 117
Alopecia (Skin and subcutaneous tissue disorders) | 62 | 58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.